CLINICAL TRIAL: NCT02520388
Title: Ph 3 Multicenter DBRCT Parallel Group Study to Evaluate Safety & Efficacy of Evening-dosed HLD200, a Novel Delayed & Extended Release Formulation (DELEXIS) of MPH HCl, on Post-waking, Early Morning Function in Children Aged 6-12 With ADHD
Brief Title: A Pivotal Efficacy Trial to Evaluate HLD200 in Children With ADHD in a Naturalistic Setting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ironshore Pharmaceuticals and Development, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLD200-108
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 5,10-dihydro-5-methylphenazine; Capsules; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HLD200 (methylphenidate) (Experimental): Experimental: HLD200 (methylphenidate)
  The investigational drug for this study is HLD200 MPH MR capsules comprised of the active pharmaceutical ingredient (MPH) in a dual-coated drug-layered core. Following a minimum 72-hour washout, subjects will be randomized (1:1) to double-blind HLD200 to be taken once daily during the evening for a period of 3-weeks prior to testing.
  Interventions: Drug: HLD200 methylphenidate hydrochloride (MPH) Capsules
- Placebo (Placebo Comparator): Placebo capsules will be composed of microcrystalline cellulose beads in place of MPH containing beads found in the HLD200 capsules. Following a minimum 72-hour washout, subjects will be randomized (1:1) to double-blind placebo to be taken once daily during the evening for a period of 3-weeks prior to testing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HLD200 methylphenidate hydrochloride (MPH) Capsules — HLD200 Doses: 40, 60 or 80 mg
  Other Names: methylphenidate
  Arms: HLD200 (methylphenidate)
Drug: Placebo
  Arms: Placebo

SUMMARY:
This Phase 3 pivotal efficacy trial will examine the effects of HLD200 (methylphenidate) in patients aged 6-12 years with ADHD in a naturalistic setting. Following a screening/washout period (Visit 1), subjects will randomized to double-blind placebo or HLD200 for a period of 3 weeks (Visits 2-5) before assessing clinical study endpoints at last study visit.

DETAILED DESCRIPTION:
To address the unmet need for early morning ADHD symptom control, Ironshore has developed a novel drug delivery system that incorporates the active ingredient methylphenidate HCl in a delayed/extended release formulation. This formulation provides a controlled, approximately 8-hour delay in initial drug release, followed by a subsequent controlled rate of drug release throughout the day. The goal of this system is to enable nighttime dosing of methylphenidate to provide control of ADHD symptoms at the beginning of the next morning (immediately upon awakening) and throughout the remainder of the day.

At Visit 2, Baseline Visit), subjects were randomized to receive either HLD200 or placebo and instructed to begin dosing at 40 mg each evening (8:00 pm ±30 minutes) for 1 week, with scheduled titration, as medically indicated and tolerated, over the subsequent 2 weeks to 60 mg (Visit 3) and 80 mg (Visit 4) and/or a dose not to exceed 3.7 mg/kg (based on the subject's most recently assessed weight). Following dose escalation above 40 mg (i.e., after Visit 3), subjects were permitted to reduce the dose by 1 step (i.e., from 60 to 40 mg or from 80 to 60 mg), if necessary, for safety or tolerability. Subjects who were unable to tolerate a dose of at least 40 mg during the final (third) week of treatment, from Visit 4 to 5, were discontinued. Subjects were also permitted to adjust the timing of the evening dosing at Visits 3 and 4 in increments of 30 to 60 minutes/week to achieve optimal morning control of observed ADHD symptoms; however, the dose was not to be taken any later than 9:30 pm or any earlier than 6:30 pm, regardless of the ±30-minute dosing window.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be male or female children (6 to 12 years at the time of consent).
2. Subjects must have a diagnosis of ADHD as defined by DSM5 criteria and confirmation using the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
3. Subjects must have a baseline ADHD-RS-IV score at or above the 90th percentile normalized for sex and age in total score. In addition, this ADHD-RS-IV total score must be ≥26 at Baseline.
4. Subjects must have a Clinical Global Impression of Severity (CGI-S) score ≥4 and a CGI-P score >10 at the Baseline Visit.
5. Subjects have demonstrated, in the judgment of the investigator, at least a partial clinical response to MPH.
6. Parental or legal guardian confirmation of the child's before-school functional impairment and/or difficulties performing a morning routine of at least 30 minutes minimum duration occurring between 6:00 and 9:00 am.
7. Subject body weight must be ≥20 kg.
8. Subject must be considered clinically appropriate for treatment with MPH and HLD200, including ability to swallow treatment capsules.
9. Subject must be in general good health based upon the medical history, physical, and laboratory examinations (including urine drug screen).
10. Subject and parent or legal guardian must be able to read, write, and/or understand at a level sufficient to provide informed consent (parent/legal guardian) and assent (subject) prior to study participation and to complete study-related materials. Subject and parent or legal guardian must plan to be available for the entire study period.
11. Female subjects of childbearing potential (i.e., post-menarche) are required to have a negative result on urine pregnancy testing at screening (and will be given specific instructions for avoiding pregnancy during the study).
12. A medically highly effective form of birth control must be used during the study and for 90 days thereafter for subjects of either sex of childbearing potential. Examples of medically highly effective forms of birth control are as follows:

    * No sexual activity
    * Use of acceptable methods of birth control including intra-uterine device, oral, implantable,or injectable contraceptives.

Exclusion Criteria:

1. History of, or current, medical condition or laboratory result which, in the opinion of the investigator, unfavorably alters the risk-benefit of study participation, may jeopardize subject safety, or may interfere with the satisfactory completion of the study and study-related procedures.
2. Serious structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, or other cardiac problems that may place the subject at increased vulnerability to the sympathomimetic effects of a stimulant drug.
3. History of seizure disorder (except febrile seizures prior to age 5 and with last occurrence at least 1 year prior to study participation), Tourette's disorder, or intellectual disability of minor severity or greater (DSM5 criteria).
4. History of psychosis, bipolar disorder, anorexia nervosa, bulimia, or suicide attempt. Current depression, anxiety, conduct/behavior disorder, substance use disorder, or other psychiatric condition which, in the investigator's opinion, may jeopardize subject safety or may interfere with the satisfactory completion of the study and study-related procedures.
5. Active suicidal ideation as evidenced by an ideation score of 2 or greater on the C-SSRS.
6. History of severe allergic reaction or intolerance to MPH.
7. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, or creatinine greater than 1.5x the upper limit of normal. Elevated bilirubin due only to Gilbert's syndrome is not exclusionary.
8. History of alcohol abuse or illicit drug use.
9. Use of prescription medications (except per protocol allowed medications) within 7 days of Baseline (Visit 2), except for ADHD stimulant medication (72 hours) and monoamine oxidase inhibitors (MAOIs) (14 days), and over-the-counter medications (except birth control and allowed medications) within the 3 days preceding Baseline (Visit 2). Medications not covered in allowed medications or prohibited medications must be cleared by the medical monitor prior to enrolling the subject.
10. Use of psychotropic medications including antidepressants, mood stabilizers, and antipsychotics.
11. Participation in a clinical trial with an investigational drug within the 30 days preceding study enrollment.
12. Previous treatment experience with HLD200.
13. Positive screening for illicit drug use or nicotine and/or current health conditions or use of medications that might confound the results of the study or increase risk to the subject.
14. In the opinion of the investigator, the subject may have problems complying with the protocol or the procedures of the protocol, or for which the study could pose unnecessary safety risks. This includes current health conditions or use of medications that might confound the results of the study or increase risk to the subject.
15. A sibling or step-sibling that is concurrently participating in this study who resides with and is cared for by the same parent/legal guardian as the subject.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Newcorn Jeffrey, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (21):
- United States (21):
  - AVIDA, Newport Beach, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - QPS MRA, dba Miami Research Associates, LLC, South Miami, Florida
  - Children's Developmental Center, P.A., Winter Park, Florida
  - Pedia Research, LLC, Owensboro, Kentucky
  - Duke University Medical Center, Duke Child and Family Study Center, Durham, North Carolina
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Bayou City Research, Ltd, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Westex Clinical Investigations, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Ericksen Research and Development, Clinton, Utah
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Storebo OJ, Storm MRO, Pereira Ribeiro J, Skoog M, Groth C, Callesen HE, Schaug JP, Darling P, Huus CL, Zwi M, Kirubakaran R, Simonsen E, Gluud C. Methylphenidate for children and adolescents with attention deficit hyperactivity disorder (ADHD). Cochrane Database Syst Rev. 2025 Dec 4;12(12):CD009885. doi: 10.1002/14651858.CD009885.pub4. PMID 41342306
- [Derived] Storebo OJ, Storm MRO, Pereira Ribeiro J, Skoog M, Groth C, Callesen HE, Schaug JP, Darling Rasmussen P, Huus CL, Zwi M, Kirubakaran R, Simonsen E, Gluud C. Methylphenidate for children and adolescents with attention deficit hyperactivity disorder (ADHD). Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD009885. doi: 10.1002/14651858.CD009885.pub3. PMID 36971690
- [Derived] Wilens TE, Faraone SV, Hammerness PG, Pliszka SR, Uchida CL, DeSousa NJ, Sallee FR, Incledon B, Newcorn JH. Clinically Meaningful Improvements in Early Morning and Late Afternoon/Evening Functional Impairment in Children with ADHD Treated with Delayed-Release and Extended-Release Methylphenidate. J Atten Disord. 2022 Mar;26(5):696-705. doi: 10.1177/10870547211020073. Epub 2021 Jun 4. PMID 34085581
- [Derived] Lopez FA, Faraone SV, Newcorn JH, Doll HA, Rhoten S, Lewis HB, Khan TF, DeSousa NJ, Sallee FR, Incledon B. Effect of Delayed-Release and Extended-Release Methylphenidate on Caregiver Strain and Validation of Psychometric Properties of the Caregiver Strain Questionnaire: Results from a Phase 3 Trial in Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2021 Apr;31(3):179-186. doi: 10.1089/cap.2020.0159. Epub 2021 Apr 1. PMID 33797983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 22 sites in the United States. First subject enrolled was on 13 August, 2015 and last subject completed was on 13 May, 2016.
Pre-assignment Details: In total, 163 particpants were enrolled in the study (completed the Baseline Visit).
Groups:
- HLD200 (Methylphenidate): Participantas recieved HLD200 capsules (containing beads with methylphenidate in a dual-coated drug-layered core; 40, 60 or 80 mg) orally once daily in the evening for 3 weeks.
- Placebo: Participants recieved placebo (matched to HLD200 capsules, but containing microcrystalline cellulose beads in place of methylphenidate) orally once daily in the evening for 3 weeks.
Period: Overall Study
Arm/Group | HLD200 (Methylphenidate) | Placebo
Started | 82 | 81
Treated | 81 | 80
Completed | 73 | 65
Not Completed | 9 | 16
Not completed — Physician Decision | 1 | 0
Not completed — Subject or parent/guardian request | 0 | 6
Not completed — Adverse Event | 1 | 4
Not completed — Lost to Follow-up | 3 | 2
Not completed — Other (reason not defined) | 4 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat
Groups:
- HLD200 (Methylphenidate): At the start of the Randomized Placebo-controlled Test Phase (Visit 2), subjects were randomized to receive either HLD200 or placebo. Subjects instructed to begin dosing at 40mg each evening (8:00 pm ±30 minutes) for 1 week, with scheduled titration, as medically indicated and tolerated, over the subsequent 2 weeks to 60 mg (Visit 3) and 80 mg (Visit 4) and/or a dose not to exceed 3.7 mg/kg (based on the subject's most recently assessed weight). Following dose escalation above 40 mg (i.e., after Visit 3), subjects were permitted to reduce the dose by 1 step (i.e., from 60 to 40 mg or from 80 to 60 mg) if necessary for safety or tolerability. Subjects who were unable to tolerate a dose of at least 40 mg during the final (third) week of treatment, from Visit 4 to 5, were discontinued. Subjects were also permitted to adjust the timing of the evening dosing at Visits 3 and 4 in increments of 30 to 60 minutes/week to achieve optimal morning control of observed ADHD symptoms; however, the dose was not to be taken any later than 9:30 pm or any earlier than 6:30 pm, regardless of the ±30-minute dosing window.
- Placebo: At the start of the randomized placebo-controlled Test Phase (Visit 2), subjects were randomized to receive either HLD200 or placebo. Placebo capsules were colour and weight matched to the active HLD200 capsules.
  Subjects instructed to begin dosing at 40mg each evening (8:00 pm ±30 minutes) for 1 week, with scheduled titration, as medically indicated and tolerated, over the subsequent 2 weeks to 60 mg (Visit 3) and 80 mg (Visit 4) and/or a dose not to exceed 3.7 mg/kg (based on the subject's most recently assessed weight). Following dose escalation above 40 mg (i.e., after Visit 3), subjects were permitted to reduce the dose by 1 step (i.e., from 60 to 40 mg or from 80 to 60 mg) if necessary for safety or tolerability. Subjects who were unable to tolerate a dose of at least 40 mg during the final (third) week of treatment, from Visit 4 to 5, were discontinued. Subjects were also permitted to adjust the timing of the evening dosing at Visits 3 and 4 in increments of 30 to 60 minutes/week to achieve optimal morning control of observed ADHD symptoms; however, the dose was not to be taken any later than 9:30 pm or any earlier than 6:30 pm, regardless of the ±30-minute dosing window.
- Total: Total of all reporting groups
Arm/Group | HLD200 (Methylphenidate) | Placebo | Total
Number analyzed (Participants) | 81 | 80 | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.6 (1.79) | 9.0 (1.73) | 9.3 (1.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 55 | 58 | 113

OUTCOME MEASURES:

1. Primary Outcome: Attention Deficit Hyperactivity Disorder Rating Scale Based on DSM-IV Criteria (ADHD-RS-IV) Total Score.
Description: The ADHD-RS-IV was developed to measure the behaviors of children with ADHD (DuPaul et al., 1998). The scale consists of 18 items designed to reflect current symptomatology of ADHD. Each item is scored in a range from 0 (reflecting no symptoms or a frequency of never or rarely) to 3 (reflecting severe symptoms or a frequency of almost always), with a range of total scores ranging from 0 to 54. In this study, a site clinican (required to be an MD, PhD, DO, licensed social worker, or any trained mental health professional approved by the sponsor) completed ADHD-RS-IV assessments at each visit using a structured interview format.
Time Frame: Last week of 3-week treatment period assessed at Visit 5.
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: ADHD-RS-IV total score
Arm/Group | HLD200 (Methylphenidate) | Placebo
Number analyzed (Participants) | 78 | 67
ADHD-RS-IV total score | 24.1 (1.5) | 31.2 (1.6)
Statistical Analysis 1: Comparison: HLD200 (Methylphenidate) vs Placebo; Test type: Superiority; p = 0.05, Mixed model repeated measures analysis

2. Secondary Outcome: Before School Functioning Questionnaire (BSFQ) Total Score
Description: The BSFQ was developed as a hybrid measure completed by a clinician or parent/legal guardian to assess commonly reported areas of morning dysfunction - both behaviors and functions associated with the post-waking, early morning period (from approximately 6:00 am to 9:00 am) - in children and adolescents with ADHD (Wilens et al., 2010; Wilens et al., 2013). Symptom severity and functional impairment were rated from 0 (none) to 3 (severe - different from peers all days, all settings) with total scores ranging from 0 to 60. Ratings were completed by a site clinician (MD, PhD, DO, licensed social worker, or trained mental health professional approved by the sponsor) at Visits 2 through 5 using a structured interview format.
Time Frame: Last week of 3-week treatment period assessed at Visit 5.
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: BSFQ total score
Arm/Group | HLD200 (Methylphenidate) | Placebo
Number analyzed (Participants) | 78 | 67
BSFQ total score | 18.7 (1.63) | 28.4 (1.73)
Statistical Analysis 1: Comparison: HLD200 (Methylphenidate) vs Placebo; Test type: Superiority; p = 0.05, Mixed model repeated measures analysis

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from the start of study treatment up to the safety follow-up assessment (35 days)
Description: Assessment of adverse events by study staff occurred at every study visit and were recorded based on spontaneous reports from subjects/parents regardless of causality. However, sleep-related adverse event were directly solicited from subjects/parents by study staff using a structured interview format to assess sleep disturbance (including sleep onset, quality and quantity), rather than obtained from spontaneous reporting.
Arm/Group | HLD200 (Methylphenidate) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/80
Other Adverse Events (participants affected / at risk) | 27/81 | 24/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HLD200 (Methylphenidate) (N=81) | Placebo (N=80)
Any Insomnia (Psychiatric disorders) | 27 | 7 — Includes: Initial insomnia, Middle insomnia, Terminal insomnia and Insomnia, not specified.
Affect lability/mood swings (Psychiatric disorders) | 5 | 1 — Combined term includes both Affect lability and Mood swings
Decreased appetite (Metabolism and nutrition disorders) | 15 | 3
Headache (Nervous system disorders) | 8 | 4
Psychomotor hyperactivity (Nervous system disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 7 | 0
Nausea (Gastrointestinal disorders) | 5 | 0
Sleep disorder (Psychiatric disorders) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No